CLINICAL TRIAL: NCT00045669
Title: A Phase 2 Study Of Imatinib Mesylate In Adenoid Cystic, Lymphoepithelioma-Like And Myoepithelial Salivary Gland Carcinomas
Brief Title: Imatinib Mesylate in Treating Patients With Salivary Gland Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000257029; PMH-PHL-009 (Other: Princess Margaret Cancer Centre); NCI-5663 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Head and Neck Cancer
Keywords: recurrent salivary gland cancer; salivary gland adenoid cystic carcinoma; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms | interventions — Imatinib Mesylate

ARMS (1):
- Imatinib Mesylate (Experimental): Adult patients with unresectable or metastatic adenoid cystic carcinoma measurable by Response Evaluation Criteria in Solid Tumors Group criteria and expressing c-kit by immunohistochemistry were treated with imatinib 400 mg orally bid. Response was assessed every 8 weeks
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have unresectable and/or metastatic salivary gland cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of imatinib mesylate, in terms of objective response rates (partial and complete responses) and duration of overall response, in patients with unresectable and/or metastatic adenoid cystic, lymphoepithelioma-like, or myoepithelial salivary gland cancer.
* Determine the safety and tolerability of this drug in these patients.
* Correlate the activity of c-kit and downstream kinases in pre- and post-treatment tumoral biopsies with clinical course in patients treated with this drug.
* Determine the effect of treatment with this drug on tumor samples from these patients in terms of proliferation, apoptosis, and angiogenesis.
* Correlate the steady state levels of this drug achieved with clinical and laboratory correlative endpoints in these patients.
* Determine whether early changes in metabolic activity correlate with molecular changes and predict outcome to therapy in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate twice daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with stable disease receive treatment for up to 6 months.

Patients are followed within 3 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 6-19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenoid cystic, lymphoepithelioma-like, or myoepithelial salivary gland cancer

  * Unresectable AND/OR
  * Radiologically documented metastatic disease
* c-kit positive tumor (1+, 2+, or 3+)
* At least 1 unidimensionally measurable lesion

  * More than 20 mm by conventional techniques OR
  * More than 10 mm by spiral CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3

Hepatic

* Bilirubin less than 1.25 times upper limit of normal (ULN)
* AST/ALT less than 2.5 times ULN

Renal

* Creatinine less than 1.25 times ULN OR
* Creatinine clearance greater than 50 mL/min

Cardiovascular

* No myocardial infarction within the past 6 months
* No congestive heart failure
* No unstable angina
* No active cardiomyopathy
* No unstable ventricular arrhythmias
* No uncontrolled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study
* No other active malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or non-melanomatous skin cancer
* No uncontrolled psychotic disorders
* No serious infections
* No active peptic ulcer disease
* No other serious medical condition that would preclude study
* No prior allergy to compounds of similar chemical or biologic composition as imatinib mesylate

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent filgrastim (G-CSF)

Chemotherapy

* At least 4 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy to sites of measurable disease

Surgery

* At least 4 weeks since prior surgery and recovered

Other

* No other concurrent investigational agents
* No concurrent therapeutic warfarin

  * Mini-dose warfarin for prophylaxis or low-molecular weight heparin allowed
* No concurrent erythromycin
* No concurrent acetaminophen doses exceeding 3 g/day

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-07; Primary Completion 2004-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George P. Browman, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre
Locations (15):
- United States (14):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - LaGrange Memorial Hospital, LaGrange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Siteman Cancer Center, St Louis, Missouri
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Hotte SJ, Winquist EW, Lamont E, MacKenzie M, Vokes E, Chen EX, Brown S, Pond GR, Murgo A, Siu LL. Imatinib mesylate in patients with adenoid cystic cancers of the salivary glands expressing c-kit: a Princess Margaret Hospital phase II consortium study. J Clin Oncol. 2005 Jan 20;23(3):585-90. doi: 10.1200/JCO.2005.06.125. PMID 15659505